CLINICAL TRIAL: NCT00876317
Title: Efficacy and Safety of Etoricoxib in Acute Soft Tissue Rheumatism Affecting the Shoulder
Brief Title: Etoricoxib in Acute Soft Tissue Rheumatism Affecting the Shoulder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Change in current areas of research interest of the collaborator
Sponsor: Clinica Virgen Milagrosa (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dr. Luis Vidal, Rheumatology, Clinica Virgen Milagrosa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36459
Record Dates: First submitted 2009-04-02; First posted 2009-04-06 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Soft Tissue Injuries of the Shoulder; Tenosynovitis and Bursitis Affecting the Shoulder
Keywords: Tenosynovitis; Bursitis
MeSH Terms: conditions — Tenosynovitis; Bursitis | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Etoricoxib 60 mg per oz for 14 days
  Interventions: Drug: Etoricoxib 60 mg
- 2 (Active Comparator): Etoricoxib 90 mg per oz for 14 days
  Interventions: Drug: Etoricoxib 90 mg

INTERVENTIONS:
Drug: Etoricoxib 60 mg — Etoricoxib 60 mg per oz per day for 14 days
  Arms: 1
Drug: Etoricoxib 90 mg — Etoricoxib 90 mg per oz for 14 days
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety two oral doses of etoricoxib (60 mg and 90 mg) daily in acute soft tissue rheumatism affecting the shoulder.

DETAILED DESCRIPTION:
The main objective of this clinical trial is the assessment of the efficacy and safety of two single daily oral doses of etoricoxib 60 mg and 90 mg over a period of 14 days in the treatment of patients with acute soft tissue rheumatism affecting the shoulder. The study will be performed according to a randomised, double blind, double-dummy, and parallel-group.

In this study we will include 300 male or female out-patients, aged 18 years or above, with acute episodes of soft tissue rheumatism affecting the shoulder (less than 5 days). The main inclusion criteria will be: Shoulder pain of acute onset of non-traumatic origin, a history of painless unrestricted motion of the affected joint immediately before the acute attack, acute one-sided shoulder pain caused by soft tissue rheumatism, patient-assessed pain on active movement exceeding 50 mm on a 100-mm visual analogue scale and symptoms requiring therapy with NSAIDs.

The main exclusion criteria will be: Active or recurrent peptic (gastric or duodenal) ulcer, history of peptic ulcer or gastrointestinal bleeding, history of other bleeding disorders other than gastro-intestinal, concomitant treatment with anti-coagulants, lithium, other NSAIDs (including aspirin doses > 150 mg) or corticosteroids, local injections of steroids in the affecting shoulder (six months previous), presence of any form of crystal, destructive, infectious or inflammatory arthropathy, osteonecrosis, previous shoulder surgery in the affected side, adhesive capsulitis, cervical radiculopathy, severe renal, cardiac or hepatic failure, uncontrolled hypertension, pregnancy or breast feeding, confined to bed, planned hospital stays or surgical procedures during the trial, planned surgical intervention of the affected shoulder during the trial, alcohol or drug abuse and inability to comply with the protocol.

The study will have 4 Visits, at Day 1 (Visit 1), at Day 3 (Visit 2), at Day 7 (Visit 3) and at Day 14 (Visit 4). Potentially eligible patients will be screened at Visit 1. Patients found to be eligible will be allocated to one of the two treatments (etoricoxib 60 mg or 90 mg). Each patient will be treated for 14 days. Early termination of study on Visit 3 (Day 7) will be possible in case of complete resolution of the symptoms. All procedures of the study must be done after the patient sign the informed consent. An ultrasound and X-ray evaluation of the affected shoulder will be done on Day 1 and haematological and biochemistry laboratory evaluation will be done on Day 1 and at the end of treatment.

The primary end-point for efficacy will be the patient's assessment of pain on active movement on Day 3, the secondary end-point(s) for efficacy will be: Patient's assessment of pain on active movement during the last 24 hours, patient's assessment of pain at rest, the Brief Pain Inventory, final global assessment of efficacy by patient at the end of the treatment, final global assessment of efficacy by investigator at the end of the treatment, withdrawal due to inadequate efficacy, patient's status (change in painful condition at the end of therapy) and paracetamol consumption used as rescue medication. The secondary end-point(s) for safety and tolerability will be: Incidence and intensity of adverse events, final global assessment of tolerability by patient, final global assessment of tolerability by investigator, incidence of laboratory-related adverse events, and withdrawal of patients due to adverse events.

The results will be tabulated and the analysis of the data will perform in order to evaluate if the efficacy of the same doses of etoricoxib (60 mg and 90 mg) are equally effective for the treatment of acute shoulder pain syndrome due to soft tissue rheumatism affecting the shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain of acute onset of non-traumatic origin (less than 5 days).
* A history of painless unrestricted motion of the affected joint immediately before the acute attack.
* Acute one-sided shoulder pain caused by soft tissue rheumatism affecting the shoulder (bicipital tendinitis, rotator cuff tendinitis or subacromial bursitis) diagnosed by clinical signs and symptoms and confirmed by ultrasound evaluation.
* Patient-assessed pain on active movement exceeding 50 mm on a 100-mm visual analogue scale.
* Symptoms requiring therapy with NSAIDs.

Exclusion Criteria:

* Active or recurrent peptic (gastric or duodenal) ulcer.
* History of peptic ulcer or gastrointestinal bleeding.
* History of other bleeding disorders other than gastro-intestinal (e.g. cerebrovascular).
* Concomitant treatment with anti-coagulants (including heparin, ticlopidine, etc.), lithium, other NSAIDs (including aspirin doses > 150 mg) or corticosteroids.
* Local injections of steroids in the affecting shoulder (within six months prior to the trial and during the trial).
* Presence of any form of crystal arthropathy (e.g. gout, pseudogout), destructive arthropathies (e.g. Charcot joints), infectious arthritis, chronic sepsis, osteonecrosis, rheumatoid inflammatory disease, previous
* shoulder surgery in the affected side, adhesive capsulitis in the affected side or cervical radiculopathy.
* Severe renal, cardiac or hepatic failure.
* Uncontrolled hypertension.
* Pregnancy or breast feeding.
* Confined to bed.
* Planned hospital stays or surgical procedures during the trial.
* Planned surgical intervention of the affected shoulder during the trial.
* Known alcohol or drug abuse.
* Inability to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pain on active movement | Day 3

SECONDARY OUTCOMES:
Brief Pain Inventory | Days 0, 3, 7 and 14
Global tolerability evaluation by the physician at the end of the study | Day 14
Incidence and intensity of adverse events | Days 3, 7 and 14
Global tolerability evaluation by the patient at the end of the study | Day 14
Evaluation of pain at resting in the affecting shoulder the last 24 hours (VAS) | Days 0, 3, 7 and 14
Pain on active movement | Day 0, 7, 14
Patient's assessment of pain on active movement during the last 24 hours | Day 0, 3, 7 and 14
Final global assessment of efficacy by patient at the end of the treatment | Day 14
Final global assessment of efficacy by investigator at the end of the treatment | Day 14
Withdrawal due to inadequate efficacy | Day 14
Paracetamol consumption used as rescue medication | Days 3, 7 and 14
Withdrawal of patients due to adverse events | Days 3, 7 and 14
Additional visits to a physician due to adverse event | Days 3, 7 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Vidal, MD, Principal Investigator — Centro Diagnóstico de la Osteoporosis y Enfermedades Reumáticas
Locations (1):
- Clínica Virgen Milagrosa, Lima, Lima Province, Peru